CLINICAL TRIAL: NCT02070328
Title: Registry Study for Proton Therapy Clinical Outcomes and Long-Term Follow-up
Acronym: Registry
Status: Recruiting | Type: Observational
Sponsor: Center for Biomedical Research, LLC (Other)
Collaborators: Provision Center for Proton Therapy (Other)
Responsible Party: Sponsor
Other Study IDs: PRO 0425
Record Dates: First submitted 2014-01-14; First posted 2014-02-25 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Proton Therapy; Registry
MeSH Terms: conditions — Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation therapy Registry: Cancer patients who have received proton therapy
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry

SUMMARY:
Proton therapy is a limited medical resource that is more expensive than conventional x-ray therapy. To correctly measure the success of proton therapy in treating different conditions, it is important to check a patient's health status after their treatment is finished. Checking on the progress of patients over many years (called long-term follow-up) is needed because the long-term effects of proton therapy are not well known.

DETAILED DESCRIPTION:
The objective of this research protocol is the development of a national Proton Therapy Center Registry for the purpose of:

1. Performing retrospective research studies on diseases treated with proton therapy throughout the United States.
2. Maintaining regular, lifetime contact with subjects in order to obtain current identification , contact information, and self/parent-reported health status in order to obtain a better understanding of overall treatment strategies and patient benefits of treatment.
3. Permitting review of medical record information contained within the Registry to identify subjects who may be eligible for participation in future research studies conducted at the Proton Therapy Institution where the participant was treated. Obtaining the permission of Research Registry participants to be contacted to ascertain their interest in participating in future research studies being conducted at their participating Proton Therapy Institution for which it appears (i.e., based on medical information contained within the Research Registry) they may be eligible.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who are receiving or seeking medical care at the participating Proton Therapy Center will be invited to participate in the Research Registry.

Exclusion Criteria:

* Subjects who do not agree to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are seen/treated at proton therapy centers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-12; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Long-term follow-up | 6 months
  Maintaining regular, lifetime contact with subjects in order to obtain current identification , contact information, and self/parent-reported health status in order to obtain a better understanding of overall treatment strategies and patient benefits of treatment.

SECONDARY OUTCOMES:
Future Research Possibilities | 12 months
  Performing retrospective research studies on diseases treated with proton therapy throughout the United States.
  Permitting review of medical record information contained within the Registry to identify subjects who may be eligible for participation in future research studies conducted at the Proton Therapy Institution where the participant was treated. Obtaining the permission of Research Registry participants to be contacted to ascertain their interest in participating in future research studies being conducted at their participating Proton Therapy Institution for which it appears (i.e., based on medical information contained within the Research Registry) they may be eligible.

CONTACTS AND LOCATIONS:
Overall Officials: James R Gray, M.D., Principal Investigator — Provision Center for Proton Therapy
Locations (3):
- United States (3):
  - Ackerman Cancer Center, Jacksonville, Florida
  - Provision CARES Proton Therapy Nashville, Franklin, Tennessee
  - Texas Center for Proton Therapy, Irving, Texas

REFERENCES:
- See also: Provision Center for Proton Therapy — http://provisionproton.com